CLINICAL TRIAL: NCT03645850
Title: Evaluation of the Efficacy and Safety of Vismed® Gel Multi 0.3% Versus Vismed® Multi 0.18% on the Treatment of Moderate to Severe Ocular Dryness
Brief Title: Evaluation of Efficacy and Safety of Vismed Gel Multi 0.3% Versus Vismed Multi 0.18% on Treatment of Ocular Dryness
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Horus Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17E4554; 2018-A01711-54 (Other: ANSM)
Record Dates: First submitted 2018-08-22; First posted 2018-08-24 (Actual); Last update posted 2018-08-24 (Actual); Status verified 2018-08

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: Parallel Assignment Because the comparator will be in commercial packaging, the blinding of the subject is not possible.
  However, the study will be blinded for the investigator: evaluations will be done by an independent investigator, different than the person who will distribute the product. Subjects will be identified by a patient number. Each patient number will be associated to a treatment number, according to a randomization list provided before the beginning of the clinical investigation, and randomized either in one of both treatment groups (Vismed Gel Multi 3% or Vismed Multi 0.18%).
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Investig. device:Vismed Gel Multi 0.3% (Experimental): Vismed gel Multi 0.3% eye drops: 1 to 2 drops in each eye between 4 and 6 times per day during 84 days
  Interventions: Device: Vismed gel Multi 0.3% eye drops
- Comparative device: Vismed Multi 0.18% (Active Comparator): Vismed Multi 0.18% eye drops: 1 to 2 drops in each eye between 4 and 6 times per day during 84 days
  Interventions: Device: Vismed Multi 0.18% eye drops

INTERVENTIONS:
Device: Vismed gel Multi 0.3% eye drops — Ophthalmic use. Vismed gel Multi 0.3% eye drops. One to two drops instilled in each eye from 4 to 6 times per day during 84 days of treatment.
  Arms: Investig. device:Vismed Gel Multi 0.3%
Device: Vismed Multi 0.18% eye drops — Ophthalmic use. One to two drops instilled in each eye from 4 to 6 times per day during 84 days of treatment.
  Arms: Comparative device: Vismed Multi 0.18%

SUMMARY:
This study is a multicentric, comparative, randomized, investigator-blinded, parallel group study to demonstrate the non-inferiority of Vismed® Gel Multi 0.3% in comparison with Vismed® Multi 0.18% in terms of cornea and conjunctiva staining (Oxford score) on patients with moderate to severe ocular dryness, after 35 days of treatment.

DETAILED DESCRIPTION:
Evaluation of the non-inferiority of Vismed® Gel Multi 0.3% in comparison with Vismed® Multi 0.18%, in terms of cornea and conjunctiva staining (Oxford score), on worse eye, between Day 0 and Day 35.

Evaluation of the non-inferiority of Vismed® Gel Multi 0.3% in comparison with Vismed® Multi 0.18%, in terms of cornea and conjunctiva staining (Oxford score), on worse eye, between Day 0 and Day 35.

* Comparison of Day 35 versus Day 0 and Day 84 versus Day 0 for each product and comparison between products for the following parameters:

  * Evolution of cornea and conjunctiva staining (Oxford score) on worse eye.
  * Evolution of DEQ-5 score (5-items Dry Eye Questionnaire).
  * Evolution of Van Bijsterveld score (Lissamine green staining) in worse eye.
  * Evolution of Schirmer test result in worse eye.
  * Evolution of Tear film Break-Up Time (TBUT) in worse eye.
  * Evolution of ocular dryness severity by evaluation of each main symptom by the patient and total score of all symptoms
  * Evaluation of treatment performance by the investigator and the patient.
* Evaluation of the average frequency of use over 84 days for both products.

ELIGIBILITY:
Inclusion Criteria:

* Sex: male or female.
* Age: more than 18 years.
* Subject with a moderate to severe dry eye syndrome needing artificial tears in the 3 months preceding the inclusion.
* Subject having used only artificial tears without preservative (NaCl 0.9%, Hydrabak®) during 1 to 2 weeks before inclusion (up to 6 times a day).
* Subject with a score ≥ 6 for the 5-Item Dry Eye Questionnaire (DEQ-5)
* Subject with at least one eye with:

  * Global ocular staining (cornea and conjunctiva) ≥4 and ≤9 on the Oxford scale (0 to 15)

AND one of the following criteria:

* Schirmer test ≥ 3 mm/5 min and ≤ 9 mm/5 min OR
* Sum of 3 measurements of Tear film Break-Up Time (TBUT) ≤ 30s.

  * Subject, having given freely and expressly his/her informed consent.
  * Subject who is able to comply with the study requirements, as defined in the present CIP, at the Investigator's appreciation.
  * In France: subject being affiliated to a health social security system. Female subjects of childbearing potential should use a medically accepted contraceptive regimen since at least 12 weeks before the beginning of the study, during all the study and at least 1 month after the study end.

Exclusion Criteria:

* Pregnant or nursing woman or planning a pregnancy during the study.
* Subject deprived of freedom by administrative or legal decision.
* Subject in a social or health institution
* Subject who is under guardianship or who is not able to express his/her consent.
* Subject being in an exclusion period for a previous study.
* Subject suspected to be non-compliant according to the Investigator's judgment.
* Subject wearing contact lenses during the study.
* Far best corrected visual acuity < 1/10
* Subject with severe ocular dryness with one of these conditions:

  * Eyelid or blinking malfunction
  * Corneal disorders not related to dry eye syndrome
  * Ocular metaplasia
  * Filamentous keratitis
  * Corneal neovascularization
* Subject with severe meibomian gland dysfunction (MGD)
* History of ocular trauma, infection or inflammation, not related to dry eye syndrome within the last 3 months prior to the inclusion.
* History of ocular allergy or ocular herpes within the last 12 months.
* Subjects who underwent ocular surgery, including laser surgery, in either eye within the last 6 months.
* Any troubles of the ocular surface not related to dry eye syndrome.
* Subject having used artificial tears in the 6 hours preceding the inclusion visit.
* Use of the following ocular treatments: isotretinoïd, cyclosporine, tacrolimus, sirolimus, pimecrolimus, punctual plugs during the month preceding the inclusion.
* Subjects who have received ocular therapy (either eye) with any ophthalmic medication, except tear substitutes, within 2 weeks prior to study start or expected to receive ocular therapy during the study.
* Any not stabilised systemic treatment, which can have an effect on performance or safety criteria, at the investigator appreciation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-09-01 (Estimated); Primary Completion 2019-03-01 (Estimated); Study Completion 2019-06-15 (Estimated)

PRIMARY OUTCOMES:
Demonstrate the non-inferiority of Vismed® Gel Multi 0.3% in comparison with Vismed® Multi 0.18% in terms of cornea and conjunctiva staining (Oxford score) on patients with moderate to severe ocular dryness, after 35 days of treatment. | 35 days
  Assess the ocular surface fluorescein staining score- mean change from Baseline in the study at D35 in ocular surface fluorescein stainig score according to a scale from zero to 15
To assess the total ocular surface fluorescein staining score at D84 | 0 and 84 days
  Mean change from Baseline (D0) in the study eye and D84 in the total ocular surface fluoresceine staining score
Evolution of DEQ-5 score | 35 days
  Evolution from Baseline of DEQ-5 questionnaire scores at day 35
Evolution of DEQ-5 score | 84 days
  Evolution from Baseline of DEQ-5 questionnaire scores at day 84
Evolution of Van Bijterveld score ( lissamine green staining) | 35 Days
  Mean change from Baseline ( D0) and D 35 in the total Van Bijterveld score
Evolution of Van Bijterveld score ( lissamine green staining) | 84 days
  Mean change from Baseline ( D0) and D 84 in the total Van Bijterveld score
Volume tear fluid secretion as assessed by schirmer test | 35 days
  Mean change from Baseline ( D0) in Volume tear fluid secretion as assessed
Volume tear fluid secretion as assessed by schirmer test | 84 days
  Mean change from Baseline ( D0) in Volume tear fluid secretion as assessed
Evolution of Tear film Break-Up Time | 35 days
  Mean change from Baseline (D0) in the study eye in TFBUT at Day 35
Evolution of Tear film Break-Up Time | 84 days
  Mean change from Baseline (D0) in the study eye in TFBUT at Day 84
Global sum score of dry eye symptoms at visit 3 - mean change from Baseline at visit 3 ( D35) | 35 days
  Mean change from Baseline in the global sum score of dry eye symptoms at D35 : discomfort,burning, stinging,eye dryness sensation, itching,foreign body sensation,photophobia, blurred vision.Each graded from 0 to 10
Global sum score of dry eye symptoms at visit 4 - mean change from Baseline at visit 3 ( D84) | 84 days
  Mean change from Baseline in the global sum score of dry eye symptoms at D84 : discomfort,burning, stinging,eye dryness sensation, itching,foreign body sensation,photophobia, blurred vision.Each graded from 0 to 10
Global treatment performance score assessed by the investigator at visit 3 | 35 days
  Total Treatment performance score graded from 0 to 4
Global treatment performance score assessed by the investigator at visit 4 | 84 days
  Total Treatment performance score graded from 0 to 4
Global treatment performance score assessed by the patient at visit 3 | 35 days
  Total Treatment performance score graded from 0 to 4
Global treatment performance score assessed by the patient at visit 4 | 84 days
  Total Treatment performance score graded from 0 to 4

CONTACTS AND LOCATIONS:
Overall Officials: Béatrice Cochener-Lamard, Prof, Principal Investigator — Hôpital Morvan, Brest, France

IPD SHARING:
Plan to Share IPD: Undecided
Depending on any journal publication of the results